CLINICAL TRIAL: NCT06258096
Title: Photobiomodulation Therapy, a Novel Approach for the Management of Taste Disorders in Cancer Patients
Brief Title: LI-TASTE Study: Light for Taste
Acronym: LI-TASTE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NL84772.018.23
Record Dates: First submitted 2024-01-30; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma
Keywords: Stemcell transplant; Light therapy; Taste changes; Dysgeusia
MeSH Terms: conditions — Multiple Myeloma; Dysgeusia

STUDY DESIGN:
Intervention Model Description: Double-blind RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation therapy (PBMT) (Experimental): Patients will receive either PBMT or sham-PBMT during admission to the hospital. The oral cavity of the patients will be exposed to LED light using a new intra-oral device on the THOR Control Unit at the intensity of 50mW/m2 for 60 seconds per dose. Additionally, the perioral region will be exposed to LED light using an extra-oral device on the THOR Control Unit at the intensity of 50mW/m2 for 60 seconds per dose.
  Interventions: Device: LX2.3 Laser and LED Photobiomodulation System
- Sham-PBMT (Sham Comparator): Patients will receive either PBMT or sham-PBMT during admission to the hospital. The sham-PBMT is the placebo treatment and consists of light of the same colour (white light with a red filter), applied in the same way as in the experimental group.
  Interventions: Device: LX2.3 Laser and LED Photobiomodulation System Sham-PBMT Setting

INTERVENTIONS:
Device: LX2.3 Laser and LED Photobiomodulation System — The LX2.3 Laser and LED Photobiomodulation system by THOR Photomedicine Ltd is a CE marked product and has a long track record of safety, usability, and effectiveness.
  Other Names: THOR Oral LED
  Arms: Photobiomodulation therapy (PBMT)
Device: LX2.3 Laser and LED Photobiomodulation System Sham-PBMT Setting — The sham setting consists of light of the same colour (white light with a red filter), applied in the same way as in the experimental group.
  Other Names: THOR Oral LED Sham Setting
  Arms: Sham-PBMT

SUMMARY:
Rationale: In 2020, 115,000 Dutch patients were diagnosed with cancer. Up to 85% of patients treated with radiotherapy involving the head and neck, chemotherapy or stem-celltransplantation (SCT) suffer from taste disorders (dysgeusia). Dysgeusia is one of the most distressing adverse effects of cancer therapy, may be long-lasting and may contribute to malnutrition and decreased QoL. Dysgeusia pathobiology is complex and relates to direct damage to taste buds by anticancer therapies, neuropathy and/or mucosal infection and inflammation. Hyposalivation and concurrent medications may also play a role as well as smoking and poor oral health. Zinc suppletion, clonazepam and delta-9-tetrahydrocannabionol have only limited success. Thus, dysgeusia in cancer patients represents a significant unmet clinical need.

Photobiomodulation therapy (PBMT) using specific wavelengths of red/near infrared light reduces oxidative stress and increases ATP in cells, which improves cell metabolism and reduces inflammation. PBMT is safe and effective for the prevention of oral mucositis and is linked to pain reduction, nerve damage recovery and improved wound healing. There is emerging evidence for PBMT to improve taste, likely based on its regenerative effects on taste buds and nerves involved in taste function. However, there is need for more reliable data on the effect of PBMT on taste. Objective: Assess the efficacy of PBMT to prevent/ameliorate dysgeusia in patients with multiple myeloma treated in Amsterdam UMC with conditioning chemo(radio)therapy followed by autologous stem-cell-transplantation.

Study design: Single centre, prospective, longitudinal, double-blinded, randomized, controlled study. Study population: Recipients of autologous hematopoietic stem cell transplantation (SCT) for the treatment of multiple myeloma in Amsterdam UMC. Intervention: Patients will be blinded to receive either PBMT or sham-PBMT. Main study parameters/endpoints: Objective and subjective taste function and taste associated covariables and their impact on QoL will be assessed.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The application of PBMT to the (peri)oral region is safe and comes with no relevant side effects. The application of PBMT or sham-PBMT will take about 10-15 minutes per treatment. The measurements at the start of the study and at the visit six weeks after SCT will last about 30 minutes. Scoring the PROMS (2 questionnaires of 1-5 questions) during hospitalization will take about five minutes per day; 2 questionnaires (30+15+ 5 questions), 10 minutes, weekly. Patients do not need to come to the hospital specifically for the study, as they already have an appointment in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a haematological malignancy
* > 18 years of age
* Receiving HDM followed by SCT
* Able and willing to give informed consent

Exclusion Criteria:

* Having taste disorders not related to SCT (e.g. COVID-19)
* History of a head and neck tumor treated with surgery and/or (chemo)radiation
* Neurological diseases (e.g. Parkinson's disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-02-29 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Objectively scored taste changes | 6 weeks
  The Medisense test will be used to assess objective taste: The ODOFIN taste strips are a validated research procedure for determining taste sensitivity. The patient's task is to choose one of the following answers: 1. Sweet, 2. Sour, 3. Salty, 4. Bitter, 5. Umami, 6. No taste. The maximum number of points is 4 points per taste.
Subjectively scored taste changes | 6 weeks
  The CiTAS-NL questionnaire will be used to assess subjective taste: Decline in basic tastes: Add up the scores of questions 2 to 6 and divide by 5. Discomfort: Add up the scores of questions 13 to 18 and divide by 6. Phantogeusia or parageusia: Add up the scores of questions 10 to 12 and divide by 3. General taste changes: Add up the scores of question 1 and from 7 to 9 and divide by 4. Overall score: Add up the scores from question 1 to 18 and divide by 18. Interpretation of score: A score lower than 6 is not significant, 6-10 indicates mild, 10-14 indicates moderate, and 15-20 indicates severe taste changes.

SECONDARY OUTCOMES:
Salivary flow | 6 weeks
  the presence and severity of hyposalivation following SCT
Xerostomia | 6 weeks
  the presence and severity of xerostomia following SCT
Oral mucositis | 6 weeks
  the presence and severity of patient reported oral mucositis following SCT
Caloric intake | 6 weeks
  the caloric intake before and after SCT
Global-health-related QoL | 3 weeks
  Global Qol will be assessed by EORTC QLQ-C30 (Version 3.0)
Oral-health-related QoL | 3 weeks
  Oral-health related QoL will be assessed by EORTC QLQ - OH15

IPD SHARING:
Plan to Share IPD: No